CLINICAL TRIAL: NCT03741101
Title: Treatment of NF1-related Plexiform Neurofibroma With Trametinib; a Single Arm, Open-label Trial With the Goals of Volumetric Partial Remission and Pain Relief
Brief Title: Treatment of NF1-related Plexiform Neurofibroma With Trametinib
Acronym: plexifpc
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUS2018-1; 2018-001846-32 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Neurofibromatosis 1; Child; Neurofibroma, Plexiform
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm study (Experimental): children treated with trametinib
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — treatment
  Other Names: mekinist

SUMMARY:
This trial, Treatment of NF1-related plexiform neurofibroma with trametinib; a single arm,open-label study with the goals of volumetric partial remission and pain relief (EudraCT 2018-001846-32, Sponsor protocol number BUS2018-1, related Novartis reference number CTMT212ASE01T) is a pediatric clinical trial that investigates the potential use of the drug trametinib (Mekinist®) as treatment for symptomatic or likely to become symptomatic NF1-related plexiform neurofibromas (PN) in children between 1 year and 17 year and 11 months of age.

Trametinib is orally administered qd at 0.025 mg/kg up to a maximum of 2 mg from six years of age and 0.032mg/kilo up to 5 years of age, provided either as tablets or as oral solution. It is manufactured and distributed by Novartis under the trade name Mekinist®.

The primary endpoint is remission of tumor volume ≥20%, evaluated using volumetric MRI at 18 and 30 months of treatment.

The secondary endpoint is reversal of pain from NF1-related PN, evaluated monthly with agespecific pain scales; VAS scale (from 8 years) or Faces Pain Scale (from 3 to 8 years).

As an exploratory measure, the potential effects of the treatment on the cognitive function will be assessed using well-established tests such as WISC-V (age range 6:0 - 16:11), NEPSY-II (age range 3:0-16:11), and CPT-3 (age range 8:0 - adult).

Cognitive dysfunction is well described in patients with NF1, and the MAPK/ERK-pathway has been indicated to be involved in cognition.

ELIGIBILITY:
Inclusion Criteria

* NF1-related PN with severe - or with high suspicion of becoming severe - manifestations
* Informed consent provided
* Age 1:0-17:11

Exclusion Criteria

* NF1-related PN does not fulfill characteristics for acceptable volumetric MRI assessments as outlined under Criteria for volumetric assessment.
* Lactating or pregnant females. Sexually active females, who do not (agree to) use safe contraception or adhere to regular controls during study. Sexually active males who do not (agree to) use a condom during coitus.
* A history of other malignancies than classic NF1-related WHO grade 1 tumors (i.e. PN or optic pathway glioma).
* A history of NF-1 related cerebral vascular anomalies (such as Moyamoya).
* Active pharmaceutical therapy for optic pathway malignancy/ies.
* Any medication for treatment of left ventricular systolic dysfunction.
* Use of any investigational drug within 30 days of the first dose of this study treatment.
* Impaired renal function (GFR under 45 ml/min/1,73m2 - It is only required to analyze eGFR if creatine is above institutional reference value for corresponding age group).
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug or excipients that contraindicate their participation.
* Active liver or biliary disease or moderate or severe liver impairment. If there are signs of liver disease (such as an increased prothrombin time or elevated transaminases),grading of the liver impairment has to be done in consultation with a hepatologist, since there is no universal definition.
* A history of hepatic sinusoid obstructive syndrome (venoocclusive disease) within the last 3 months.
* A history of heparin-induced thrombocytopenia.
* A history of interstitial lung disease or pneumonitis.
* A history of retinal vein occlusion (RVO).
* A history of Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection. Subjects with a confirmed cleared HBV and HCV infection may be enrolled.
* Presence of a condition that will interfere significantly with the absorption of drugs.
* Evidence of cardiovascular risk, such as left ventricular ejection fraction (LVEF) below the lower limit of normal (LLN), a corrected QT-interval (Qtc) >480 milliseconds, clinically significant uncontrolled arrhythmia, congestive heart failure, or acute coronary syndrome or history thereof.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Remission of tumor volume ≥20% | 0 - 30 months.
  Final and primary analysis of primary outcome measure - of pooled data at 30 months (end of study) with volumetric mri of tumor volume versus volume at enrolment.
Remission of tumor volume ≥20% | 0 - 18 months
  Interim analysis of pooled data at 18 months with volumetric mri of tumor volume versus volume at enrolment. This is an interim analysis of primary outcome and not primary analysis of primary outcome".

SECONDARY OUTCOMES:
Reversal of NF1-related PN elicited - VAS scale pain | 0 - 30 months.
  Evaluated with monthly VAS pain scale from 8 years at enrolment. Monthly. 0-10 point scale. Descriptive. Analysis of pooled data after month 30.
Reversal of NF1-related PN elicited pain - Faces Pain Scale | 0 - 30 months.
  Evaluated with monthly Faces Pain Scale from under 8 years at enrolment. Monthly. 0-10 scale. Descriptive. Analysis of pooled data after month 30.

OTHER OUTCOMES:
Cognitive performance. Exploratory. WISC V. | 0-18 months.
  Change of full scale IQ or primary indexes of WISC V. Pooled data after 18 months versus before/at enrolment; with p-value <0.05.
Cognitive performance. Exploratory. NEPSYII. | 0-18 months.
  Change of Learning and Memory functions and visuospatial functions, pooled data after 18 months versus before/at enrolment (selected test from NEPSYII,; with p-value <0.05.
Cognitive performance. Exploratory. CPT3. | 0-18 months.
  Change in attention, pooled data after 18 months versus before/at enrolment (CPT-3); with p-value <0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Sigurdsson, Principal Investigator — Skane University Hospital
Locations (1):
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical trial register EU — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2018-001846-32